CLINICAL TRIAL: NCT03191968
Title: A Pilot, Randomized Controlled Trial Adding Behavioral Counseling to Supervised Physical Activity in Prostate Cancer Survivors
Brief Title: Prostate Cancer Survivors and Exercise and Behavioral Counseling
Acronym: BOOST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2017-04

CONDITIONS: Physical Activity; Cancer of the Prostate; Cognitive Impairment; Quality of Life
Keywords: Behavior change; Prostate cancer; Behavioral counseling; Physical Activity; Randomized controlled trial
MeSH Terms: conditions — Motor Activity; Prostatic Neoplasms; Cognitive Dysfunction | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised PA Plus Behavioral Counseling (Experimental): 25 prostate cancer survivors will receive supervised physical activity and behavioral counseling (SPA+BC) based on the M-PAC. In addition to supervised physical activity, behavioral counseling sessions will be delivered with a PA specialist based on the Multi-process Action Control (M-PAC) framework and include behavior change techniques addressing information regarding the consequences, social support, goal setting, self-monitoring, cues and prompts, barrier identification, intention formation, planning, and habit and identity formation
  Interventions: Behavioral: Supervised Physical Activity Plus Behavioral Counseling
- Supervised PA Plus Exercise Counseling (Active Comparator): 25 prostate cancer survivors will supervised physical activity and exercise counseling (SPA+EC).In addition to the supervised exercise sessions, standard exercise counseling will be delivered by a PA specialist to teach proper PA and resistance training techniques, how to monitor intensity, and to progress PA safely and effectively to achieve the public health PA guideline.
  Interventions: Behavioral: Supervised Physical Activity Plus Exercise Counseling

INTERVENTIONS:
Behavioral: Supervised Physical Activity Plus Behavioral Counseling — In addition to supervised physical activity, behavioral counseling sessions will be delivered with a PA specialist based on the Multi-process Action Control (M-PAC) framework and include behavior change techniques addressing information regarding the consequences, social support, goal setting, self-monitoring, cues and prompts, barrier identification, intention formation, planning, and habit and identity formation
  Arms: Supervised PA Plus Behavioral Counseling
Behavioral: Supervised Physical Activity Plus Exercise Counseling — In addition to the supervised exercise sessions, standard exercise counseling will be delivered by a PA specialist to teach proper PA and resistance training techniques, how to monitor intensity, and to progress PA safely and effectively to achieve the public health PA guideline.
  Arms: Supervised PA Plus Exercise Counseling

SUMMARY:
This study will evaluate the feasibility of delivering a supervised physical activity program plus standard exercise counseling (SPA+EC) versus a supervised physical activity plus motivationally-enhanced behavioral counseling (SPA+BC) in prostate cancer survivors (PCS). Fifty participants (n=25) will be randomized to receiving SPA+EC or SPA+BC (n=25). We hypothesize that PCS receiving the SPA+BC intervention will result in greater increases in objectively-assessed physical activity compared with PCS receiving the SPA+EC intervention.

DETAILED DESCRIPTION:
Physical activity (PA) has a positive impact on clinical outcomes such as improvement in overall QoL, cancer-specific mortality, reducing treatment-related toxicities, and reducing fatigue across many cancer survivor groups including PCS. Despite these benefits of regular PA, the majority of PCS are still not meeting public health PA guidelines.

Short-term supervised PA programs have been shown to improve health-related fitness and patient-reported outcomes in PCS, but PA declines significantly after the supervised intervention has been completed. Research examining the effect of short- term supervised exercise programs on motivational outcomes and longer term PA among cancer survivors is limited, especially theoretical approaches to identify key motivational outcomes for behavior change.

This study will pilot a two-armed, single blind, RCT comparing SPA+EC to SPA+BC. The proposed RCT in PCS is noteworthy given that it differs from standard approaches to supervised PA with the addition of a behavioral counseling component. This rigorous comparison condition will provide further evidence that theoretically-informed interventions are needed to adopt long-term PA maintenance.

The program's supervised exercise length will be 6 weeks, followed by a tapered contact throughout the a 6-week home-based component through 'booster' behavioral counseling delivered via telephone. In terms of study measures, objective measures of PA will be used (i.e.,accelerometry, inclinometers), and cardiorespiratory fitness will be evaluated using maximal graded exercise testing via treadmill. Additional secondary outcomes include cognitive function, quality of life, physical function, body composition, motivational outcomes, sexual functioning, masculinity, sedentary behavior, and cardiorespiratory fitness.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years and older
* Histologically confirmed prostate cancer (Stage I-IIIa) but now cured or in remission
* Ability and willingness to effectively communicate in English
* Not meeting physical activity guidelines of ≥150 minutes of vigorous physical activity

Exclusion Criteria:

* Severe coronary artery disease (Canadian Cardiovascular Society class III or greater)
* Significant congestive heart failure (New York Heart Association class III or greater)
* Uncontrolled pain
* Neurological or musculoskeletal co-morbidity inhibiting exercise
* Diagnosed psychotic, addictive or major cognitive disorders
* Absent for more than 3 consecutive days during the 12-week intervention
* High risk individuals (i.e., men who have symptomatic and known cardiovascular, pulmonary and/or metabolic disease) as determined by the risk stratification questionnaire

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Objectively assessed physical activity | Change in from baseline at 12 weeks
  Objective Physical activity will be measured using an activity device, accelerometry (i.e., Actigraph GTX3+)

SECONDARY OUTCOMES:
Self-reported physical activity | Change in from baseline at 12 weeks
  Self-reported physical activity will be assessed using the Godin Leisure-Time Exercise Questionnaire
Physical Function | Change in from baseline at 12 weeks
  Mobility-related fitness parameters will be measured through the six-items of the Seniors' Fitness Test.
General quality of life | Change in from baseline at 12 weeks
  Self-reported quality of life measured via the Functional Assessment of Cancer Therapy (FACT-G) for general quality of life.
Prostate-specific quality of life | Change in from baseline at 12 weeks
  Self-reported quality of life measured via the FACT-Prostate for prostate-specific quality of life.
Cancer-related fatigue | Change in from baseline at 12 weeks
  Self-reported fatigue will be assessed using the FACT-Fatigue
General well-being | Change in from baseline at 12 weeks
  Self-reported Short-Form 36 will be used for assessing general well-being.
Body composition | Change in from baseline at 12 weeks
  Body composition will be estimated using anthropometric measurements will be taken - height, weight and waist circumference.
Cardiorespiratory fitness | Change in from baseline at 12 weeks
  Aerobic endurance capacity will be assessed by using the modified Balke sub-maximual exercise test.
Cognitive function | Change in from baseline at 12 weeks
  The primary set of neuropsychological assessments will be assessed using the validated NIH Toolbox Cognition Battery. This battery consists of tests to assess Executive Function, Attention, Episodic Memory, Language, Processing Speed and Working Memory.
Sexual Health | Change in from baseline at 12 weeks
  The International Index of Erectile Function (IIEF) will be used to assess sexual health including erectile function, orgasmic function, sexual desire, intercourse satisfaction and overall satisfaction.
Relationship quality | Change in from baseline at 12 weeks
  The Perceived Relationship Quality Components (PRQC) Inventory will be used to assess relationship quality.
Masculine self-esteem | Change in from baseline at 12 weeks
  Masculine self-esteem will be assessed using the Masculinity in Chronic Disease Inventory (MCD-I).
Motivational outcomes | Change in from baseline at 12 weeks
  multi-process action control (M-PAC) framework assessing attitudes, subjective norms, perceived behavioral control, planning, habit, and identity
Self-reported sedentary behavior | Change in from baseline at 12 weeks
  sitting time as measured by via self-report using the Measuring Older Adults' Sedentary Time (MOST) questionnaire which assesses sitting while watching TV, using the computer, hobbies, socializing, transportation, doing hobbies, and other activities.
Objectively assessed sedentary behavior | Change in from baseline at 12 weeks
  Objective measures of sitting time will be assessed using an activity device, inclinometers (i.e., ActivPALs)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Trinh, PhD, Principal Investigator — University of Illinois at Urbana-Champaign; Edward McAuley, PhD, Study Director — University of Illinois at Urbana-Champaign; Art F Kramer, PhD, Study Director — University of Illinois at Urbana-Champaign and Northeastern University; Kendrith M Rowland, MD, Study Director — Carle Cancer Center
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Courneya KS, Friedenreich CM, Reid RD, Gelmon K, Mackey JR, Ladha AB, Proulx C, Vallance JK, Segal RJ. Predictors of follow-up exercise behavior 6 months after a randomized trial of exercise training during breast cancer chemotherapy. Breast Cancer Res Treat. 2009 Mar;114(1):179-87. doi: 10.1007/s10549-008-9987-3. Epub 2008 Apr 4. PMID 18389368
- [Background] Keogh JW, MacLeod RD. Body composition, physical fitness, functional performance, quality of life, and fatigue benefits of exercise for prostate cancer patients: a systematic review. J Pain Symptom Manage. 2012 Jan;43(1):96-110. doi: 10.1016/j.jpainsymman.2011.03.006. Epub 2011 Jun 2. PMID 21640547
- [Background] Mishra SI, Scherer RW, Geigle PM, Berlanstein DR, Topaloglu O, Gotay CC, Snyder C. Exercise interventions on health-related quality of life for cancer survivors. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD007566. doi: 10.1002/14651858.CD007566.pub2. PMID 22895961
- [Background] Antonelli J, Freedland SJ, Jones LW. Exercise therapy across the prostate cancer continuum. Prostate Cancer Prostatic Dis. 2009;12(2):110-5. doi: 10.1038/pcan.2009.4. Epub 2009 Mar 10. PMID 19274062
- [Background] Bonn SE, Sjolander A, Lagerros YT, Wiklund F, Stattin P, Holmberg E, Gronberg H, Balter K. Physical activity and survival among men diagnosed with prostate cancer. Cancer Epidemiol Biomarkers Prev. 2015 Jan;24(1):57-64. doi: 10.1158/1055-9965.EPI-14-0707. Epub 2014 Dec 19. PMID 25527697
- [Background] Rock CL, Doyle C, Demark-Wahnefried W, Meyerhardt J, Courneya KS, Schwartz AL, Bandera EV, Hamilton KK, Grant B, McCullough M, Byers T, Gansler T. Nutrition and physical activity guidelines for cancer survivors. CA Cancer J Clin. 2012 Jul-Aug;62(4):243-74. doi: 10.3322/caac.21142. Epub 2012 Apr 26. PMID 22539238
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Baumann FT, Zopf EM, Bloch W. Clinical exercise interventions in prostate cancer patients--a systematic review of randomized controlled trials. Support Care Cancer. 2012 Feb;20(2):221-33. doi: 10.1007/s00520-011-1271-0. Epub 2011 Oct 12. PMID 21989678
- [Background] Courneya KS, Segal RJ, Gelmon K, Reid RD, Mackey JR, Friedenreich CM, Proulx C, Lane K, Ladha AB, Vallance JK, McKenzie DC. Predictors of supervised exercise adherence during breast cancer chemotherapy. Med Sci Sports Exerc. 2008 Jun;40(6):1180-7. doi: 10.1249/MSS.0b013e318168da45. PMID 18460985
- [Background] Trinh L, Plotnikoff RC, Rhodes RE, North S, Courneya KS. Feasibility and preliminary efficacy of adding behavioral counseling to supervised physical activity in kidney cancer survivors: a randomized controlled trial. Cancer Nurs. 2014 Sep-Oct;37(5):E8-22. doi: 10.1097/NCC.0b013e3182a40fb6. PMID 24232192
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Treanor CJ, Li J, Donnelly M. Cognitive impairment among prostate cancer patients: An overview of reviews. Eur J Cancer Care (Engl). 2017 Nov;26(6). doi: 10.1111/ecc.12642. Epub 2017 Feb 7. PMID 28169490
- [Derived] Trinh L, Kramer AF, Rowland K, Strom DA, Wong JN, McAuley E. A pilot feasibility randomized controlled trial adding behavioral counseling to supervised physical activity in prostate cancer survivors: behavior change in prostate cancer survivors trial (BOOST). J Behav Med. 2021 Apr;44(2):172-186. doi: 10.1007/s10865-020-00185-8. Epub 2020 Sep 26. PMID 32979134